CLINICAL TRIAL: NCT01386320
Title: A Randomised, Blinded Comparison of an Ultrasound Guided Ankle Block Compared to a Nerve Stimulator Guided Ankle Block for Pain Relief After Forefoot Surgery.
Brief Title: Ultrasound Guided Ankle Block Versus Medial Forefoot Block for Forefoot Surgery
Acronym: USGAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R0929 10/1304/1
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pain Relief After Forefoot Surgery
Keywords: anaesthetic techniques, regional; surgery orthopaedic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided ankle block (Active Comparator): Subjects in this arm will be given an ultrasound guided ankle block prior to foot surgery.
  Interventions: Procedure: Ultrasound guided ankle block
- Medial forefoot block (Active Comparator): Subjects in this arm will be given a nerve-stimulator guided forefoot block prior to anaesthesia and forefoot surgery
  Interventions: Procedure: Medial forefoot block

INTERVENTIONS:
Procedure: Ultrasound guided ankle block — Under ultrasound guidance, block of the tibial nerve, superficial and deep branches of the common peroneal nerve and saphenous nerves will be carried out using 12 mls 0.5% levobupivacaine and 12 mls 0.75% levobupivacaine.
  Arms: Ultrasound guided ankle block
Procedure: Medial forefoot block — Using peripheral nerve stimulator guidance, the tibial and common peroneal nerves will be blocked ( plus the saphenous nerve ), using a total of 12 mls 0.75% levobupivacaine and 12 mls 0.5% levobupivacaine.
  Arms: Medial forefoot block

SUMMARY:
Forefoot surgery includes bunion surgery and similar reconstructive bone cutting surgery and is very painful. Local anaesthetic nerve blocks have been used for many years to help alleviate pain following this surgery. The present study aims to compare a new ultrasound guided nerve block to a well established nerve stimulator guided technique. Comparisons will include time taken to carry out the block, speed of onset of numbness and duration and quality of pain relief after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Fit adult patients requiring forefoot surgery with bone cutting.

Exclusion Criteria:

* Morbid obesity (BMI >40), known contraindications to regional anaesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time taken to carry out each local anaesthetic block | Over forty five minutes from the start of the study.
  Time taken between opening sterile packs and completion of local anaesthetic block is measured by a blind observer.

SECONDARY OUTCOMES:
Onset of local anaesthesia | Over thirty minutes from completion of the local anaesthetic block.
  Following administration of the local block, development of anaesthesia will be measured looking at cold and pin-prick sensation by a blind observer.
Duration of pain relief following local anaesthetic block. | Over 24 hours following surgery.
  Pain relief will be assessed over 24 hours following surgery, to assess its duration and quality, by a blind observer.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Coe, FRCA, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Castle Hill Hospital, Castle Road, Cottingham, Hull, East Yorkshire, United Kingdom